CLINICAL TRIAL: NCT02281370
Title: A Phase I, Open-label, Randomized, Three-period Cross-over Study Evaluating the Effect of Cyclosporine on the Pharmacokinetics of Eltrombopag in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of Eltrombopag and Cyclosporine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201583
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: cyclosporine; drug-drug interaction; pharmacokinetics; eltrombopag; SB-497115
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SEQUENCE D0, D1, D2 (Experimental): Participants will receive treatment D0 in treatment period 1, D1 in treatment period 2 and D2 in treatment period 3 (one treatment per period). Where D0=eltrombopag 50 milligram (mg), D1= cyclosporine 200 mg + eltrombopag 50 mg, and D2= cyclosporine 600 mg + eltrombopag 50 mg. Treatment periods will be separated by washout periods of 3-10 days
  Interventions: Drug: Eltrombopag; Drug: Cyclosporine
- SEQUENCE D1, D0, D2 (Experimental): Participants will receive treatment D1 in treatment period 1, D0 in treatment period 2 and D2 in treatment period 3 (one treatment per period). Where D0=eltrombopag 50 mg, D1= cyclosporine 200 mg + eltrombopag 50 mg, and D2= cyclosporine 600 mg + eltrombopag 50 mg. Treatment periods will be separated by washout periods of 3-10 days
  Interventions: Drug: Eltrombopag; Drug: Cyclosporine
- SEQUENCE D1, D2, D0 (Experimental): Participants will receive treatment D1 in treatment period 1, D2 in treatment period 2 and D0 in treatment period 3 (one treatment per period). Where D0=eltrombopag 50 mg, D1= cyclosporine 200 mg + eltrombopag 50 mg, and D2= cyclosporine 600 mg + eltrombopag 50 mg. Treatment periods will be separated by washout periods of 3-10 days
  Interventions: Drug: Eltrombopag; Drug: Cyclosporine

INTERVENTIONS:
Drug: Eltrombopag — White to off white bi-convex round tablets containing eltrombopag 50 mg for oral administration
Drug: Cyclosporine — Soft gelatine capsule containing cyclosporine 100 mg for oral administration. Cyclosporine will be administered at the doses of 200 mg (2 x 100 mg capsules) or 600 mg (6 x 100 mg capsules)

SUMMARY:
A drug-drug interaction study between eltrombopag and cyclosporine is being conducted to support the use of these drugs together in subjects, such as those with severe aplastic anemia or immune thrombocytopenia purpura. The primary objective of the study is to evaluate the effect of cyclosporine on the pharmacokinetics of eltrombopag. This is a Phase I, open-label, randomized, three-period cross-over study in healthy adult subjects. The study consists of a screening visit and three treatment periods. All subjects will be randomized to receive one of the three treatments in each treatment period separated by washout periods of 3-10 days. The total duration of a subject's participation in the study from screening to final discharge is up to approximately 6 weeks (assuming 3 day washouts between treatment periods). Approximately 39 healthy subjects will be enrolled with the goal of completing at least 10 subjects per sequence (total 30).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 64 years of age inclusive.
* Healthy subjects.
* Body weight >=60 kilograms (kg) for men and women and body mass index (BMI) within the range 24.7-32.0 kg/meter squared (m^2) inclusive.
* Male: Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception during the study.
* Female of non-child bearing potential.
* Female of child-bearing potential who has a negative serum or urine pregnancy test and is willing to practice acceptable methods of birth control during the study.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected (QTc) > 450 millisecond (msec): The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read.

For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used.

* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days.
* Requiring the use of oral or injectable strong Cytochrome P3A4 (CYP3A4) and Breast cancer resistance protein (BRCP) inhibitors or use of other CYP3A4 and BCRP inhibitors/inducers within 14 days prior to dosing.
* History of regular alcohol consumption within 1 month of the study.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products within 30 days prior to screening.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Platelet counts or creatinine levels that exceed the upper limit of the normal range.
* Presence of hepatitis B surface antigen (HBsAg) or presence of hepatitis B core antibody (HBcAb), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment - A positive pre-study drug/alcohol screen.
* A positive test for human immune virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* The subject has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2014-12-24 (Actual); Study Completion 2014-12-24 (Actual)

PRIMARY OUTCOMES:
Plasma eltrombopag area under time-concentration curve from time zero to infinity (AUC[0-inf]) | Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose in each treatment period
Plasma eltrombopag maximum observed concentration (Cmax) | Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose in each treatment period

SECONDARY OUTCOMES:
Composite of plasma eltrombopag pharmacokinetic (PK) parameters | Pre-dose and at 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, and 72 hours post-dose in each treatment period
  PK parameters include: area under time-concentration curve from time zero to the time of last quantifiable concentration (AUC[0-t]), the percentage of AUC(0-inf) obtained by extrapolation (%AUCex), time to occurrence of Cmax (tmax), terminal phase half-life (t1/2), and apparent oral clearance (CL/F)
Vital signs assessment | Up to 6 weeks
  Vital signs will include temperature, systolic and diastolic blood pressure, pulse rate, and respiratory rate
Composite clinical laboratory assessments including hematology, clinical chemistry and urinalysis parameters | Up to 6 weeks
Number of participants with adverse events (AEs) | From the start of study treatment until the end of treatment period 3 (assessed up to 18 days)
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Electrocardiogram (ECG) assessment | Up to 6 weeks
  Single 12-lead ECG will be obtained following eltrombopag dosing using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT interval (QTc)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Aslanis V, Zhang J, Lomeli B, Grosch K, Ouatas T. Effect of cyclosporine coadministration on the pharmacokinetics of eltrombopag in healthy volunteers. Cancer Chemother Pharmacol. 2018 Nov;82(5):847-855. doi: 10.1007/s00280-018-3677-6. Epub 2018 Aug 31. PMID 30171280
- See also: Results for study 201583 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/201583?search=study&search_terms=201583#rs